CLINICAL TRIAL: NCT02453958
Title: Non-Invasive Assay to Discriminate Mild Traumatic Brain Injury
Brief Title: Mild Traumatic Brain Injury Discrimination
Acronym: MTBID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Empirical Technologies Corporation (Industry)
Collaborators: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency); Walter Reed Army Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: ETC_mTBI_001
Record Dates: First submitted 2015-05-20; First posted 2015-05-27 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Brain Concussion
Keywords: Injury; Brain; Traumatic Mild; Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion; Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mTBI-diagnosed group (Experimental): Subjects diagnosed with mTBI were assessed with a multi-modal assessment system.
  Interventions: Device: Multi-modal assessment system
- non mTBI-diagnosed group (Experimental): Non-concussed subjects were assessed with a multi-modal assessment system.
  Interventions: Device: Multi-modal assessment system

INTERVENTIONS:
Device: Multi-modal assessment system — Subjects were assessed using a multi-modal concussion assessment battery incorporating eye-tracking, balance, and neurocognitive tests

SUMMARY:
Evaluation of the utility of a multi-modal assessment tool in distinguishing between individuals with and without a history of mild traumatic brain injury.

DETAILED DESCRIPTION:
This was a preliminary validational study of a multi-modal concussion assessment battery incorporating eye-tracking, balance, and neurocognitive tests on a new hardware platform, the Computerized Brain Injury Assessment System (CBIAS). Using receiver operator curve (ROC) analyses, 1) a subset of the most discriminating neuro-physiological assessment tests involving smooth pursuit eye motion (SPEM) tracking errors, corrective saccade counts, a balance score ratio sensitive to vestibular balance performance and two neurocognitive tests of response speed and memory/incidental learning, was identified, 2) the enhancement in discriminatory capability of detecting concussion-related deficits through the combination of the identified subset of assessments was demonstrated, and 3) the effectiveness of a robust and readily implemented global scoring approach was demonstrated for both eye track and balance assessment tests. These results are significant in introducing a comprehensive solution for concussion assessment that incorporates an economical, compact and mobile hardware system and an assessment battery that is multi-modal, time efficient and whose efficacy has been demonstrated on a preliminary basis. This represents a significant step toward the goal of a system capable of making a dependable return-to-play/duty determination based on concussion likelihood.

ELIGIBILITY:
Inclusion Criteria:

* Military personnel
* Age 18 to 45
* Diagnosis of mTBI within past 5 years
* Rancho Los Amigos Scale score of 7 or above

Exclusion Criteria:

* Non-military individuals
* Below age 18 or older than 45
* No diagnosis of mTBI within past 5 years
* Rancho Los Amigos Scale score of 6 or below

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Receiver-operator-curve area under the curve (AUC) | up to 5 years
  Each test's discrimination capability was quantified using AUC and p value

CONTACTS AND LOCATIONS:
Overall Officials: Martin C. Baruch, PhD, Principal Investigator — Empirical Technologies Corporation